CLINICAL TRIAL: NCT03129672
Title: Distal Tibia Sarcoma Treatment Using Allograft Arthrodesis of the Ankle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Patricia Bonilla (Other)
Collaborators: Hospital del Niño "Dr. José Renán Esquivel" (Other)
Responsible Party: Sponsor-Investigator, Patricia Bonilla, Orthopedic Oncologist MD, Hospital del Niño "Dr. José Renán Esquivel"
Organization: Hospital del Niño "Dr. José Renán Esquivel" (Other)
Other Study IDs: 000001
Record Dates: First submitted 2015-10-13; First posted 2017-04-26 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Bone Neoplasm
Keywords: allograft; distal tibia sarcoma
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: allograft arthrodesis of ankle — patients that underwent trought a block resection of a malignant tumor of the distal tibia and reconstruction with allograft arthrodesis

SUMMARY:
The study show the clinical results of limb salvage for primary malignant bone tumor of the distal tibia using block excision of the tumor and reconstruction with allograft arthrodesis with different methods of fixation (plates or intramedullary nail system)

DETAILED DESCRIPTION:
It is well known that before the 1980's the usual treatment for the sarcomas of the distal tibia was amputation (1). Currently, however, after the improvement of the chemotherapy treatments, potential reconstructions of the area in well studied patients are possible, and for that we have a wide range: auto graft, allograft and prosthetic reconstructions (2, 3)

Is important to know that osteosarcoma still meant the principal diagnosis, followed by the Ewing sarcoma and synovial sarcoma, but their malignant potency is lower than when they are present in the rest of the body (4, 5, and 6)

The purpose of this study is to recollect the patients' data followed from different institutions and countries that have the criteria for their inclusion in the study (primary malignant bone tumor of the distal tibia that underwent block excision of the tumor and reconstruction with allograft arthrodesis from the patient management for any of the multidisciplinary sarcoma team including in this study).

ELIGIBILITY:
Inclusion Criteria:

- all patients with histopathologyc diagnosis of a primary malignant bone tumor at the distal tibia that went through a tumor resection and received reconstruction with allograft as first surgical treatment

Exclusion Criteria:

* none histopatologic proved diagnosis
* patients that received other kind of surgical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients that were diagnosis with primary malignant bone tumor of the distal tibia and went trough resection and reconstruction with allograft
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-05-20 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
principal diagnosis of the patients that wen trough ankle after resection of a primary malignant tumor of the distal tibia | 1 month
  osteosarcoma: 5 patientas (2 females of 18 and 15 years old and 3 males of 19, 24 and 16 years old) telangiectasic osteosarcoma (1 female of 21 years old) Ewing sarcoma (1 male of 33 years old)

SECONDARY OUTCOMES:
mobility | 5 month to 10 years follow up
  surgical site infection, non union, malunion, osteosynthesis material failure
mortality | 5 months to 10 years follow up
  secundary of the primary tumor diagnosis or metastatic disease of it
MSTS SCORE | 5 month to 10 years follow up
  total points score of the msts score at the final follow up

CONTACTS AND LOCATIONS:
Overall Officials: patricia bonilla, MD, Principal Investigator — Hospital del Niño
Locations (1):
- Panama Children Hospital, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burrows HJ, Wilson JN, Scales JT. Excision of tumours of humerus and femur, with restoration by internal prostheses. J Bone Joint Surg Br. 1975 May;57(2):148-59. PMID 1141281
- [Background] Ebeid W, Amin S, Abdelmegid A, Refaat Y, Ghoneimy A. Reconstruction of distal tibial defects following resection of malignant tumours by pedicled vascularised fibular grafts. Acta Orthop Belg. 2007 Jun;73(3):354-9. PMID 17715726
- [Background] Liu T, Guo X, Zhang X, Li Z, Zhang Q. Reconstruction with pasteurized autograft for primary malignant bone tumor of distal tibia. Bull Cancer. 2012 Sep;99(9):87-91. doi: 10.1684/bdc.2012.1626. PMID 22863837
- [Background] Ruggieri P, Angelini A, Jorge FD, Maraldi M, Giannini S. Review of foot tumors seen in a university tumor institute. J Foot Ankle Surg. 2014 May-Jun;53(3):282-5. doi: 10.1053/j.jfas.2014.01.015. PMID 24751209
- [Background] Azevedo CP, Casanova JM, Guerra MG, Santos AL, Portela MI, Tavares PF. Tumors of the foot and ankle: a single-institution experience. J Foot Ankle Surg. 2013 Mar-Apr;52(2):147-52. doi: 10.1053/j.jfas.2012.12.004. Epub 2013 Jan 16. PMID 23333280
- [Background] Zeytoonjian T, Mankin HJ, Gebhardt MC, Hornicek FJ. Distal lower extremity sarcomas: frequency of occurrence and patient survival rate. Foot Ankle Int. 2004 May;25(5):325-30. doi: 10.1177/107110070402500509. PMID 15134614
- [Background] Clayer M, Doyle S, Sangha N, Grimer R. The toronto extremity salvage score in unoperated controls: an age, gender, and country comparison. Sarcoma. 2012;2012:717213. doi: 10.1155/2012/717213. Epub 2012 Sep 13. PMID 23028240
- [Background] Ozger H, Eralp L, Turker M, Basaran M. Surgical treatment of malignant tumors of the foot and ankle. Int J Clin Oncol. 2005 Apr;10(2):127-32. doi: 10.1007/s10147-004-0470-9. PMID 15864699
- [Background] Enneking WF, Dunham W, Gebhardt MC, Malawar M, Pritchard DJ. A system for the functional evaluation of reconstructive procedures after surgical treatment of tumors of the musculoskeletal system. Clin Orthop Relat Res. 1993 Jan;(286):241-6. PMID 8425352